CLINICAL TRIAL: NCT06730893
Title: Shared Decision-Making for Determining Treatment Strategies in Low-Risk Thyroid Cancer: a Multicenter Cluster-Randomized Controlled Trial
Brief Title: Shared Decision-Making for Determining Treatment Strategies in Low-Risk Thyroid Cancer
Acronym: MAeSTro-SDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Nowon Eulji Medical Center (Unknown); Hanyang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0008
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Cancer; Papillary Thyroid Carcinoma
Keywords: Active surveillance; Shared decision making
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SDM Group (Shared Decision-Making Group; Intervention Group) (Experimental): * Patients will receive detailed information, including an information leaflet about treatment options.
  * Clinicians will guide patients through a structured SDM protocol before finalizing the treatment decision.
  Interventions: Other: SDM protocol
- SC Group (Standard Care Group; Control Group) (No Intervention): - Patients will receive standard medical care following current clinical practices without the SDM protocol.

INTERVENTIONS:
Other: SDM protocol — Card news and Videos related to general knowledge and treatment of low-risk thyroid cancer
  Arms: SDM Group (Shared Decision-Making Group; Intervention Group)

SUMMARY:
This study is a multicenter cluster-randomized controlled trial conducted in Korea. A parallel, two-group cluster-randomized design will be used to test whether the Shared decision-making Group (SDM; intervention) is different from the Standard Care Group (SC; control).

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to evaluate whether the group provided with a decision support tool for treatment planning (Intervention; SDM group) demonstrates improved satisfaction with the decision-making process compared to the group receiving standard care (Control; SC group) among patients diagnosed with low-risk thyroid cancer who need to determine their treatment plan.

The data are collected from patients who are diagnosed with low-risk PTC and Twenty doctors with various experience of AS will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older with a thyroid nodule of 1.0 cm or less confirmed as Bethesda category V (suspicious for PTC) or VI (PTC) based on cytopathological examination, or Bethesda category III (atypia of undetermined significance) with a confirmed BRAF V600E mutation.
* Patients with no evidence of distant metastasis, cervical lymph node metastasis, recurrent laryngeal nerve invasion, or tracheal invasion. Additionally, no evidence of extrathyroidal extension (ETE) should be present, and the tumor must not belong to high-risk subtypes of PTC (e.g., diffuse sclerosing, columnar cell, or solid subtype).

Exclusion Criteria:

* Patients who cannot undergo regular follow-up or are expected to have difficulties with follow-up.
* Patients with indeterminate or benign findings on thyroid biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Decision Conflict Scale: DCS | at enrollment
  which assesses an individual's perception and understanding of decision-making by 16 items. The scale is 5-point Likert scale from 0 (Strongly Agree) to 4 (Strongly Disagree), and scores are calculated through a) summed, b) divided by 16, and c) multiplied by 25, and range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

SECONDARY OUTCOMES:
Decision Regret Scale: DRS | at 6month, 12month after enrollment
  measures distress and remorse after making a healthcare decision. Scale ranges from 1 (Strongly agree) to 5(Strongly Disagree). The final score, the items are summed and averaged. ranging from 0 (no regret) to 100 (high regret).
Shared Decision Making Questionnaire (SDM-Q-9) | at enrollment, and 6month, 12month after enrollment
  a nine-item questionnaire assessing the quality of SDM from both patient and clinician perspectives. Scale ranges from 1(completely disagree) to 6(completely agree). Higher scores are indicative of more SDM.
Patients' Perceived involvement of Care Scale (PICS) | at enrollment, and 6month, 12month after enrollment
  a 13-item questionnaire evaluating patient engagement in primary care [12]. It measures Clinician's information provision, patient's proactive information-seeking, and patient participation in treatment decisions (5-point Likert scale; 1 = Strongly Disagree, 5 = Strongly Agree). Higher scores indicate lower clinician control and greater patient involvement in decision-making.
multifocal approach to sharing in shared decision making(Mappin'SDM) | at enrollment, and 6month, 12month after enrollment
  that incorporates physician, patient, and observer perspectives during medical consultations. a 15-item tool adapted from the 12-item OPTION scale to evaluate observed patient involvement in decision-making [13]. Each item consists of behavioral and outcome components (a total of 30 items), rated by patients, clinicians, and observers (through real-time or via video review). Scale ranges from 0(not at all) to 5(absolutely true). High scores indicate high quality of decision-making communication across patient engagement.
Comparison of Quality of Life between the shared decision group and standard care group | at enrollment, and 6month, 12month after enrollment
  The Quality of Life - Thyroid (QOL-Thyroid) questionnaire was 30 items. These are assigned to four scales, each reflecting an aspect of QoL. Physical well-being is measured with two items and 13 questions, psychological well-being with 13 items and 22 questions, social concerns with eight items and 14 questions, and spiritual well-being with seven items and questions. Response options range from '0 = worst outcome' to '10 = best outcome' on an ordinal 11-point scale.
Hospital Anxiety and Depression | at enrollment, and 6month, 12month after enrollment
  a 14-item tool (7 for anxiety, 7 for depression), developed to measure hospital patients' levels of anxiety and depression. Each item is rated on a 0-3 scale, with total scores ranging from 0 to 21 per subscale. A cutoff score of 8 or higher indicates clinically significant symptoms, based on Korean validation studies.

CONTACTS AND LOCATIONS:
Overall Officials: Young Joo Park, Principal Investigator — Seoul National University Hospital; Eun Kyung Lee, Principal Investigator — National Cancer Center; Min Joo Kim, Principal Investigator — Seoul National University Bundang Hospital; Young Shin Song, Principal Investigator — SMC-SNU Boramae Medical Center; Kyong Yeun Jung, Principal Investigator — Nowon Eulji Medical Center; Shin Je Moon, Principal Investigator — Hanyang University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee EK, Kim MJ, Hwangbo Y, Moon JH, Cho SW, Chai YJ, Choi JY, Jung YS, Lee KE, Chung EJ, Kim K, Kim SJ, Kim W, Kim YH, Lee YK, Jang J, Song YS, Yi KH, Yu HW, Moon S, Jung KY, Kim HJ, Ryu CH, Ryu J, Seok J, Kang SH, Lee S, Chu AJ, Lee CY, Lee JY, Lim H, Kim JH, Park SK, Park YJ. Shared Decision-Making for Determining Treatment Strategies in Low-Risk Thyroid Cancer: Protocol of a Multicenter Cluster-Randomized Trial (MAeSTro-SDM). J Korean Med Sci. 2026 Jan 26;41(4):e58. doi: 10.3346/jkms.2026.41.e58. PMID 41589080